CLINICAL TRIAL: NCT03574025
Title: An Observational Study of Neurodevelopmental Outcome After Cardiac Arrest in Children Admitted to Paediatric Intensive Care in the United Kingdom and Ireland
Brief Title: NEUROlogical Prognosis After Cardiac Arrest in Kids
Acronym: NEUROPACK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: NEUROPACK study protocol
Record Dates: First submitted 2017-10-30; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Arrest
Keywords: Observational, Paediatric, Cardiac Arrest, PICU,
MeSH Terms: conditions — Heart Arrest | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Arrest Questionnaire: Children who will survive 3 months after Cardiac Arrest
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — To telephone the patient/family to look into how the patient is doing, moderate/severe brain damage.

SUMMARY:
Each year around 2000 children have a cardiac arrest in the United Kingdom (UK) and approximately one fifth are admitted to Pediatric Intensive Care Unit. Many of these children eventually die and among those who survive, some will be left with brain damage which could affect their quality of life. Currently, it is difficult for doctors to predict how much brain damage there is at an early stage after cardiac arrest and if this will improve in time.

NEURO-PACK aims to follow up children 3 months after their cardiac arrest to assess their quality of life and current functional status (has the child returned to usual routine as before cardiac arrest/mild disability, can the child not participate in certain activities as they were before the cardiac arrest/moderate disability, or if the child has near to no mobility/severe disability). Investigators will find this out by using a questionnaire and the research team will telephone patients and their families 3 months after the child's cardiac arrest. This telephone call should take no longer than 30 minutes. This will then be analysed and will help towards constructing a tool which will help doctors to predict which children who have had a cardiac arrest may survive with minimal brain damage.

DETAILED DESCRIPTION:
Patients will be recruited from participating PICU's. There is currently lack of accurate data to enable clinicians to predict which of these children die or survive with brain injury. This affects clear communication with families as well as decisions to apply critical care interventions by clinicians. There is also an important knowledge gap with regards to outcome of children who are admitted to pediatric intensive care after a cardiac arrest and then survive to discharge.

Inclusion Criteria:

1. Patients aged 24 hours up to 16th birthday
2. Requiring > 1minute cardiopulmonary resuscitation
3. Admitted to PICU after Out of Hospital Cardiac Arrest or In Hospital Cardiac Arrest
4. Requiring mechanical ventilation at PICU admission
5. Surviving to 3 months follow up.

Exclusion criteria:

1. Cardiac arrest occurring within a PICU or NICU (Neonatal Intensive Care Unit)
2. Clinical team at participating sites feel inclusion is inappropriate
3. Parent/ guardian or family member unable to understand the telephone questionnaires for outcome assessments in English

The NEURO-PACK observational study enables the prospective collection of a cohort of children after out-of-hospital or in-hospital cardiac arrest. Data will be collected prospectively after eligible patients are screened and informed consent has been obtained. Participants and their families will be contacted by the Trials office,3 months after the patients cardiac arrest to complete a questionnaire over the telephone regarding functional status. Only contact information of the parents/guardians will be shared with the central Trials Office once informed consent has been obtained so that follow-up assessments can be completed. This information will be stored in locked cabinets, in a swipe card Trials Office based in Birmingham for five years, in line with Good Clinical Practice (GCP) guidance.

The information collected from patients and their families will be analyzed and used to help construct a clinical prediction tool which will help clinicians to predict which children who have had cardiac arrest may survive with minimal brain damage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 24 hours up to 16th birthday
2. Requiring > 1minute cardiopulmonary resuscitation
3. Admitted to PICU after Out of Hospital Cardiac Arrest or In Hospital Cardiac Arrest
4. Requiring mechanical ventilation at PICU admission
5. Surviving to 3 months follow up.

Exclusion Criteria:

1. Cardiac arrest occurring within a PICU or NICU (Neonatal Intensive Care Unit)
2. Clinical team at participating sites feel inclusion is inappropriate
3. Parent/ guardian or family member unable to understand the telephone questionnaires for outcome assessments in English

Ages: 24 Hours to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged more than 24 hours and up to their 16th birthday who are admitted to PICU after a cardiac arrest outside of the unit.
  Patients aged less than 24 hours will not be included as these patients are frequently managed within the neonatal intensive care unit setting. Patients aged 16 years or greater are frequently managed in the UK within the adult intensive care setting. Only patient admitted to a PICU will be eligible.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Survival with good neurodevelopmental outcome assessed using the Vineland Adaptive Behavioral Score 2nd Edition (VABS-II). | 3 months after date of cardiac arrest
  The VABS-II is a measure of adaptive behavior validated from birth to adulthood. VABS-II standardized score > 70 is pre-defined as a 'Good outcome'. A score of 70 or less and death is a 'Poor outcome'. The VABS-II outcome score will be used to create a clinical prediction model of neurodevelopmental outcome within one hour of admission to pediatric intensive care for future reference that clinicians can use to predict which children with cardiac arrest may survive with minimal brain damage.

SECONDARY OUTCOMES:
Neurodevelopmental outcome assessed using the Pediatric Cerebral Performance and Category (PCPC) and Pediatric Overall Performance Category Scale (POPC) | 3 months after date of cardiac arrest
  Pediatric Cerebral Performance Category (PCPC) measures cognitive impairment after child's critical illness. Scale 1 to 6 (1 Normal, 2 Mild disability, 3, Moderate disability, 4, Severe disability, 5 Coma/vegetative state, 6, Brain death/death). Pediatric Overall Performance Category Scale (POPC).assesses functional morbidity. Scale 1 to 6 (1 Good overall performance, 2 Mild overall disability, 3 Moderate overall disability, 4 Severe overall disability, 5 Coma or vegetative state, 6 Brain death/death).

CONTACTS AND LOCATIONS:
Overall Officials: Barney Scholefield, Study Chair — Birmingham Women's and Children's Hospital
Locations (1):
- Birmingham Women and Children's Hospital PICU, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual participant data, however, we will be using and sharing data collected as a whole to construct a prediction tool to help clinicians predict the level of brain damage after cardiac arrest occurs.

REFERENCES:
- [Derived] Scholefield BR, Martin J, Penny-Thomas K, Evans S, Kool M, Parslow R, Feltbower R, Draper ES, Hiley V, Sitch AJ, Kanthimathinathan HK, Morris KP, Smith F; NEUROPACK Investigators for the Paediatric Intensive Care Society-Study Group (PICS-SG). NEUROlogical Prognosis After Cardiac Arrest in Kids (NEUROPACK) study: protocol for a prospective multicentre clinical prediction model derivation and validation study in children after cardiac arrest. BMJ Open. 2020 Sep 25;10(9):e037517. doi: 10.1136/bmjopen-2020-037517. PMID 32978195